CLINICAL TRIAL: NCT04226040
Title: Degree-of-worry and Illness Perception in Patients Suffering From Acute Illness in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Hejdi Gamst-Jensen, Principal Investigator, Hvidovre University Hospital
Other Study IDs: HvidovreDOW1
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Acute Illness
Keywords: degree-of-worry; illness perception; acute illness; emergency department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DOW and illness perception: Exploration of the association between DOW and illness perception
  Interventions: Behavioral: DOW and illness perception

INTERVENTIONS:
Behavioral: DOW and illness perception — Acutely ill patients are exposed to a survey regarding their degree of worry and illness perception

SUMMARY:
This study explores whether and how DOW, as a PRO marker, can contribute to triage in the Emergency Departments. The study is designed as a mixed-method study consisting of a survey among acutely ill patients and qualitative semi-structured interviews.

DETAILED DESCRIPTION:
In Emergency Departments (ED) in Denmark and internationally, triage manuals are used to divide incoming patients according to their acute clinical severity, and thus assess who should be examined and treated first. However, the triage manuals are criticized for being imprecise in the intermediate categories. Furthermore, the triage manuals, nationally and internationally, are criticized for not adequately involving the patient's perspective and context. In addition, triage is not independent of personal factors and workload, which may contribute to interprofessional variation. Further, patients themselves express a desire to be even more involved. Also, the relationship between patient and healthcare professional has a direct impact on the quality of health services, however, there are divergent perceptions of what patient involvement entails. Patient-Reported Outcome (PRO) data is one way in which patient involvement can occur. PRO is data reported directly from the patient without interference from the healthcare professional and is thus self-reported data, typically generated through survey studies among patients. A strength of PRO data is that these are often more sensitive which may, for example, demonstrate a higher degree of severity of the patient's symptoms. Furthermore, it is considered a strength that PRO data can be used at both group level, for example in quality assurance, as well as at an individual level to support the decision making of healthcare professionals and thereby ensure efficient use of resources. Due to lack of evidence-based knowledge in the field and despite the potential of using PRO data, the information of patients and / or relatives is not used systematically in the Emergency Department. This also applies in the acute contact, where an imprecise initial evaluation of the patient's overall medical needs can cause both over- and under-triaging to the detriment of the overall patient course. The result is an inappropriate allocation of resources at the organizational level and a poorer quality in the treatment process. This points to the need to use relevant patient-reported measures (PROM), the tool for measuring PROs. One such instrument is Degree-of-Worry (DOW), which measures the patient's self-reported level of worry. DOW is a ten-point score of self-reported worry (from 1 = minimal concern to 10 = maximally concerned), reflecting the patient's own assessment of acute illness and own perception of concern. DOW has been scientifically tested in connection with telephone triage at the medical helpline 1813 (MH1813) as a five-point score. The patient's DOW, measured at the time the patient makes his first call to the MH1813, is strongly associated with the probability of acute hospitalization within 48 hours. However, a pilot test with DOW as a five-point score in the Emergency Department indicates a ceiling effect, by which DOW will be presented as a 10-point score in this setting. DOW has the potential to increase patient safety, create greater patient involvement and increase efficiency so that the lengths of stay reflects the triage level. A previous study suggests that DOW could also be used advantageously in other similar settings, such as Emergency Department, which, however, requires that potential implementation barriers is examined.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* cognitively intact
* consent to participation.

Exclusion Criteria:

* patients arriving to the ED regarding injury
* patient with the highest triage level
* demented patients
* intoxicated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The survey: 1004 adults (≥18 years of age) who accept to participate in the study. The patients are at the Emergency Department due to acute illness.
  The interviews: of the 1004 patients 10 (+/- 10 patients are invited to participate in a semi-structured interview. The recruitment is based on purposeful sampling with maximum variation.
Sampling Method: Non-Probability Sample
Enrollment: 944 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
DOW and illness perception | 30 minutes
  Self-reported degree-of-worry during acute illness scored on a 1-10 scale (1=minimal concern, 10=maximum concern) and illness perception measured using the Brief illness perception Questionnarie

SECONDARY OUTCOMES:
DOW and re-presentation in the Emergency Department | 30 days
  Self-reported degree-of-worry during acute illness scored on a 1-10 scale (1=minimal concern, 10=maximum concern) and representation in the Emergency Department during the following 30 days
DOW and patient barriers | 30 minutes
  10 (+/- 10) semi-structured interviews to explore potential patient barriers to implement the DOW-scale in Emergency Departments

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jensen AN, Kallemose T, Frostholm L, Gamst-Jensen H. Correlation between illness perceptions and self-reported degree-of-worry in somatic ill patients in emergency care: a Danish cross-sectional study. BMJ Open. 2024 Nov 1;14(10):e089595. doi: 10.1136/bmjopen-2024-089595. PMID 39486818